CLINICAL TRIAL: NCT01618357
Title: Pre-Operative PARPi and Irradiation (POPI) in Women With an Incomplete Response to Neo-Adjuvant Chemotherapy for Breast Cancer
Brief Title: Pre-Operative Radiation and Veliparib for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Richard Zellars (Other)
Responsible Party: Sponsor-Investigator, Richard Zellars, Professor and Chairman of the Department of Radiation Oncology, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J11155; 1503214668 (Other: Indiana University IRB)
Record Dates: First submitted 2012-01-20; First posted 2012-06-13 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Veliparib; ABT-888; Radiation; POPI
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation; Mastectomy, Segmental; Mastectomy; veliparib

STUDY DESIGN:
Intervention Model Description: A dose finding trial to assess the acute and late toxicity of pre-operative PARPi and concurrent radiation in women with stage II-IV invasive breast cancer who have had an incomplete response to NAC. Our primary goal is to assess the acute toxicity a dose finding trial to assess the acute and late toxicity of pre-operative of this combined modality therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All subjects will receive pre-operative Neo-Adjuvant Chemotherapy (NAC) but only those with an incomplete response to NAC will be treated with the PARPi experimental portion of the trial explained below. Those with a complete response will be treated per standard of care.
  Interventions: Radiation: Radiation; Procedure: Lumpectomy/Mastectomy; Drug: Veliparib

INTERVENTIONS:
Radiation: Radiation — Patients will receive radiation therapy at a dose of 2.35 Gy per fraction to the breast and regional nodal region for 16 fractions to a total dose of 37.5 Gy. Treatments will be given Monday through Friday. Radiation therapy will start on day 1 of Veliparib.
Procedure: Lumpectomy/Mastectomy — Resection of breast cancer.
Drug: Veliparib — Pills to be taken twice a day during radiation and for one week after completion of radiation for a total of 29 days.

SUMMARY:
The investigators' primary aim is to determine the safety, tolerability and maximum tolerated dose (within 50 - 200mg/BID dose range) when combining veliparib and radiation.

The investigators' exploratory aim is to serially assess apoptosis/proliferation biomarkers, and gene and protein expression profiles for correlation with tumor response to POPI.

Study Plan:

It will be a standard 3+3 dose finding trial in which the MTD will be defined as the dose below the level at which >1 DLT is observed in 3-6 patients. Women with node positive disease prior to NAC and >1.0 cm residual breast disease and/or clinically positive nodal disease after NAC will be offered participation in the research phase of this study.

Women with residual disease >1cm or +/-LN after NAC (Med Onc's choice) will be offered pre-operative Veliparib and concurrent whole breast and regional nodal irradiation. Four (4) dose levels of Veliparib will be evaluated with concurrent whole breast and regional nodal irradiation (WB/RNI). The starting dose of Veliparib will be 50 mg BID, will increase in 50 mg increments to a maximum of 200 mg BID and be delivered concurrently with 235 cGy QD x 16 to the breast and SCV/Axilla.

Accrual: Up to 41 patients

DETAILED DESCRIPTION:
Neo adjuvant (Primary) chemotherapy has revolutionized the management of locally advanced breast. Two large prospective American studies have shown that NAC provides in vivo chemo-sensitivity information, and allows a greater percentage of women to have breast conserving therapy. Additionally and importantly, these two trials also showed that 20-30% of the women treated with NAC achieve a pathologic complete response (pCR) and have a better disease free and overall survival than those women who did not achieve pCR.

Unfortunately, 70-80% of patients receiving NAC do not achieve a pCR and many still must undergo a mastectomy due to an insufficient partial response. Researchers have attempted to increase the rate of pCR by adding radiation to NAC with mixed response rates. The varying rates of pCR in the above studies are likely due to the various chemotherapeutic agents used and timing of therapies yet also may represent the limitation of efficacy in combining these chemotherapy agents with radiation. What is needed is a better agent that can potentiate the effects of preoperative radiation.

One possible agent that may potentiate the effects of radiation is an inhibitor of Poly(ADP-ribose)-polymerase (PARP). PARP is a nuclear enzyme that recognizes deoxyribonucleic acid (DNA) damage and facilitates DNA repair. Cancer cells are often deficient in DNA repair. Deficiencies in DNA repair make these cancers more dependent on PARP. An inhibitor of PARP would further hamper the cancer cell's DNA repair capability. So theoretically, the efficacy of DNA damaging agents, such as radiation and chemotherapy, should be potentiated when these therapeutic modalities are combined with PARP inhibition.

Indeed, as expected, PARP inhibitors (PARPi), such as Veliparib, have been shown in pre-clinical studies to potentiate the effects of radiation and chemotherapy in several malignancies. Thus, we hypothesize that concurrent Veliparib and pre-operative breast irradiation, in women who have residual disease after NAC, will result in an increased tumor response rate. This improved tumor response will not only increase the rate of BCT, but possibly, by increasing the rate of pCRs, also improve overall survival.

However, before this hypothesis can be adequately tested, one must assess the safety of combining radiation and Veliparib. Consequently we propose a trial of Pre-Operative PARPi and Irradiation (POPI) in women with an incomplete response to NAC. It will be a standard 3+3 dose finding trial in which the MTD will be defined as the dose below the level at which >1 DLT is observed in 3-6 patients. Women with node positive disease prior to NAC and >1.0 cm residual breast disease and/or clinically positive nodal disease after NAC will be offered participation in this study. Four (4) dose levels of Veliparib will be evaluated with concurrent whole breast and regional nodal irradiation (WB/RNI). The starting dose of Veliparib will be 50 mg BID, will increase in 50 mg increments to a maximum of 200 mg BID and be delivered concurrently with 235 cGy QD x 16 to the breast and SCV/Axilla.

ELIGIBILITY:
Inclusion Criteria for Observation

* Patient must be female and 18 years of age or older.
* Patients must have histologically confirmed (by routine H&E staining) adenocarcinoma of the breast or axillary node. Patients with squamous, or metaplastic carcinomas or sarcomas of the breast are NOT eligible.
* Patient must have had a bilateral mammogram prior to NAC unless there is only one breast.
* Patient must have a Medical Oncology consult and be recommended to receive neoadjuvant chemotherapy for a stage IIB through IV carcinoma.
* Patients must not have received prior radiation therapy to the involved breast at any time for any reason due to the potential for cumulative toxicities.

Inclusion Criteria for Treatment with Veliparib and Radiation

* Patient must have a history and physical within 2 weeks prior to the start of any protocol therapy (radiation and veliparib).
* Patient must have > 1.0 cm residual in-breast cancer (via positive biopsy) or clinically positive residual nodal disease. Incident breast biopsies only permitted prior to POPI to confirm residual disease after NAC.
* Hematology:

  1. Absolute Neutrophil Count (ANC) ≥ 1000/mm3
  2. Platelet Count ≥ 100,000/mm3
  3. Hemoglobin ≥ 9.0 g/dL (after transfusion if required)
* Renal Function:

  a. Creatinine Serum ≤ 2.0 mg/dl or Creatinine Clearance ≥45mL/min
* Hepatic Function:

  1. Bilirubin ≤ 1.5 mg/dL (≤ 3.0 mg/dL with liver metastasis)
  2. Serum Glutamic-Oxaloacetic Transaminase (SGOT) ≤ 2.5 × ULN (≤ 5.0 × ULN with liver metastasis)
  3. Serum Glutamic-Pyruvic Transaminase (SGPT) ≤ 2.5 × ULN (≤ 5.0 × ULN with liver metastasis) ULN = Upper normal limit of institution's normal range
  4. If calculated creatinine clearance is < 45 mL/min, a 24-hour urine collection for creatinine clearance may be performed.
  5. Subjects with Gilbert's disease may have bilirubin up to 2.5 mg/dL (or 3.0 mg/dL with liver (metastasis).
* Patients must not be pregnant due to the potential for fetal harm as a result of this treatment regimen. Women of child-bearing potential must also have a negative pregnancy test within 2 weeks prior to start of protocol therapy (radiation and veliparib).
* Women of childbearing potential must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and up to 2 months following completion of protocol therapy

  1. Total abstinence from sexual intercourse (minimum one complete menstrual cycle)
  2. A vasectomized partner
  3. Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration
  4. Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
* Patients must not have a serious medical or psychiatric illness which prevents informed consent or compliance with treatment.
* All patients must be informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.
* Patients must have a performance status 0 or 1 by ECOG criteria (Appendix I)

Exclusion Criteria for Consent B

* Women who have a < 1.0 cm and are cN0 after NAC are not eligible.
* Last dose of chemotherapy, immunotherapy, biologic therapy, or investigational therapy, was less than 21 days prior to protocol therapy (radiation and veliparib). There are no limitations on the type or number of prior regimens. Hormonal therapy and Traztusumab are permitted during POPI.
* Bisphosphonates, hormone modification therapy, and trastuzumab are permitted without restriction.
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or prior anti-cancer treatment.
* If female, subject is pregnant or breast-feeding
* Clinically significant and uncontrolled major cardiac, respiratory, renal, hepatic, gastrointestinal, hematologic or neurological/psychiatric disease or disorder, including but not limited to:

  1. Active uncontrolled infection
  2. Symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
  3. Any other illness condition(s) that could exacerbate potential toxicities, confound safety assessments, require excluded therapy for management, or limit compliance with study requirements. Questions regarding inclusion of individual subjects should be directed to the PI.
* Unable to swallow and retain oral medications.
* History of seizure disorder.
* Known contraindication to enhanced MRI and CT, including but not limited to:

  1. Presence of metal objects within the body such as a cardiac pacemaker, implanted cardiac defibrillator, brain aneurysm clips, cochlear implant, ocular foreign body, or shrapnel.
  2. History of immediate or delayed hypersensitivity reaction or other contraindication to contrast agents including but not limited to gadolinium and iodine.
* Previous enrollment on another study involving the investigation of veliparib (ABT- 888), with the exception of receiving a single dose of study drug.
* Consideration by the Investigator, for any reason, that the subject is an unsuitable candidate to receive veliparib (ABT-888) and/or breast irradiation.

Inclusion of Underrepresented Populations Individuals of all races and ethnic groups are eligible for this trial. There is no bias towards age or race in the clinical trial outlined. This trial is open to the accrual of women only.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-07-22 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
POPI Safety, Tolerability, and MTD | 1 year
  To determine the safety, tolerability and maximum tolerated dose (within 50 - 200 mg/BID dose range) when combining Veliparib and radiation.

OTHER OUTCOMES:
Biomarkers | baseline
  Serially assess apoptosis/proliferation biomarkers via immunohistochemestry (IHC), gene microarray and proteomic analyses
Biomarkers | Cycle 1 (each cycle is 29 days)
  Serially assess apoptosis/proliferation biomarkers via immunohistochemestry (IHC), gene microarray and proteomic analyses
Biomarkers | Cycle 2 (each cycle is 29 days)
  Serially assess apoptosis/proliferation biomarkers via immunohistochemestry (IHC), gene microarray and proteomic analyses
Biomarkers | Cycle 3 (each cycle is 29 days)
  Serially assess apoptosis/proliferation biomarkers via immunohistochemestry (IHC), gene microarray and proteomic analyses
Biomarkers | Post Radiation (up to 3 months afterwards)
  Serially assess apoptosis/proliferation biomarkers via immunohistochemestry (IHC), gene microarray and proteomic analyses
Gene and protein expression | Baseline
  Create profiles for correlation with tumor response to POPI via immunohistochemestry (IHC), gene microarray and proteomic analyses
Gene and protein expression | Cycle 1 (each cycle is 29 days)
  Create profiles for correlation with tumor response to POPI via immunohistochemestry (IHC), gene microarray and proteomic analyses
Gene and protein expression | Cycle 2 (each cycle is 29 days)
  Create profiles for correlation with tumor response to POPI via immunohistochemestry (IHC), gene microarray and proteomic analyses
Gene and protein expression | Cycle 3 (each cycle is 29 days)
  Create profiles for correlation with tumor response to POPI via immunohistochemestry (IHC), gene microarray and proteomic analyses
Gene and protein expression | Post Radiation (up to 3 months afterwards)
  Create profiles for correlation with tumor response to POPI via immunohistochemestry (IHC), gene microarray and proteomic analyses

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zellars, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (6):
- United States (6):
  - I U Health West, Avon, Indiana
  - IU Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana